CLINICAL TRIAL: NCT03995160
Title: Influence of Closed Suction Drainage After Total Knee Replacement on Patient's Reported Outcome and Basic Morphology Results, and Inflammation Factors
Brief Title: Influence of Closed Suction Drainage After Total Knee Replacement.
Acronym: TKR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Artur Stolarczyk, Head of the Department of Orthopaedics and Rehabilitation, Principal Investigator, Clinical Professor, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TKR/ Warsaw MU
Record Dates: First submitted 2019-04-25; First posted 2019-06-21 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Total Knee Replacement
Keywords: total; knee; arthroplasty; tkr; drainage; haematoma
MeSH Terms: conditions — Hematoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total knee replacement with use of closed suction drainage (Active Comparator): Use of closed suction drainage following total knee replacement in treatment of knee primary osteoarthritis
  Interventions: Procedure: Use of closed suction drainage following total knee arthroplasty
- Total knee replacement without use of closed suction drainage (Active Comparator): Without the use of closed suction drainage following total knee replacement in treatment of knee primary osteoarthritis
  Interventions: Procedure: Abstain of using a closed suction drainage

INTERVENTIONS:
Procedure: Use of closed suction drainage following total knee arthroplasty — Use of closed suction drainage following total knee arthroplasty
  Other Names: Redon's drain
  Arms: Total knee replacement with use of closed suction drainage
Procedure: Abstain of using a closed suction drainage — Abstain of using a closed suction drainage following total knee arthroplasty
  Arms: Total knee replacement without use of closed suction drainage

SUMMARY:
The aim of the study will be to compare functional outcomes, basic morphology results, number of blood transfusions, costs of hospitalization, and inflammation factors, following total knee replacement (with use of one type of endoprosthesis) comparing use of closed suction drainage (CSD). Use of closed suction drainage may have influence on patients functional outcome.

DETAILED DESCRIPTION:
Patients with primary knee osteoarthritis will be included in a randomized controlled trial and assigned to total knee arthroplasty with or without closed suction drainage. Subjects will be evaluated preoperatively, 1-day, 3-, 6- and 12-month postoperatively.

Change in morphology results will be measured by comparing preoperative and postoperative levels of haematocrite, haemoglobin, erythrocytes, and platelets.

Change in the number of blood transfusions will be measured by analyzing the number of needed transfusion of packed red blood cells in the postoperative period during stay in the hospital.

Change in levels of inflammation factors will be measured by analyzing the level of C-reactive protein in first and third day postoperatively.

Change in body temperature wille be measured daily by analyzing body temperature from day of the surgery until the day of discharge from the hospital

Presence of haematoma will be evaluated daily in the postoperative period by clinical examination.

Change in Western Ontario and McMasters University Osteoarthritis Index (WOMAC) Pain Score will be measured from baseline (can be measured anytime to a maximum of one month before surgery) 3,6 and 12 months post-operatively

Change in Western Ontario and McMasters University Osteoarthritis Index (WOMAC) Function Score will be measured from baseline (can be measured anytime to a maximum of one month before surgery) 3,6 and 12 months post-operatively

Costs of hospitalization will be measured by comparing cost of hospitalization between two analyzed groups

ELIGIBILITY:
Inclusion Criteria:

* patient's consent for anticipation in the study
* arthroplasty in one knee

Exclusion Criteria:

* patient's lack of consent for anticipation in the study
* haematological diseases
* reoperations in the area of endoprosthesis
* medical history of any surgical intervention on the lower limb

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-11-02 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in haematocrite levels | from baseline (can be measured anytime to a maximum of one month before surgery) to 1-day, 3,6 and 12 months post-operatively
  Measuring results of haematocrite (in percentage in 1 ml of blood sample)
Change in the number of blood transfusions | from baseline to the 1-,2-,3- days postoperatively
  Measuring the number of needed transfusion of packed red blood cells in the postoperative period
Change in levels of inflammation factors | from baseline (can be measured anytime to a maximum of one month before surgery) to 1-day, 3,6 and 12 months post-operatively
  Measuring the level of C-reactive protein
Change in haemoglobin levels | from baseline (can be measured anytime to a maximum of one month before surgery) to 1-day, 3,6 and 12 months post-operatively
  Measuring results of haemoglobin (g/dL)
Change in erythrocytes levels | from baseline (can be measured anytime to a maximum of one month before surgery) to 1-day, 3,6 and 12 months post-operatively
  Measuring results of erythrocytes (number/ml)
Change in platelets levels | from baseline (can be measured anytime to a maximum of one month before surgery) to 1-day, 3,6 and 12 months post-operatively
  Measuring results of platelets (number/ml)

SECONDARY OUTCOMES:
Change in Western Ontario and McMasters University Osteoarthritis Index (WOMAC) Pain Score from baseline | from baseline (can be measured anytime to a maximum of one month before surgery) 3,6 and 12 months post-operatively
  The WOMAC Pain score is derived from a sub-section of the Knee injury and Osteoarthritis Outcome Score (KOOS) Knee Survey. The WOMAC Pain scores range from 0-100 with lower scores considered lower pain.
Change in Western Ontario and McMasters University Osteoarthritis Index (WOMAC) Function Score from baseline | from baseline (can be measured anytime to a maximum of one month before surgery) 3,6 and 12 months post-operatively
  The WOMAC Function score is derived from a sub-section of the Knee injury and Osteoarthritis Outcome Score (KOOS) Knee Survey. The WOMAC Function scores range from 0-100 with lower scores considered to have better function.
Change in body temperature | from baseline to the 1-,2-,3- days postoperatively
  Measuring body temperature from day of the surgery to the hospital until the day of discharge from the hospital
Influence of using CSD on costs of hospitalization | from baseline to the one year postoperatively
  Comparing cost of hospitalization between two analyzed groups

CONTACTS AND LOCATIONS:
Overall Officials: Artur Stolarczyk, MD, PhD, Study Director — Medical University of Warsaw; Marcin Wojewodzki, Principal Investigator — Medical University of Warsaw

IPD SHARING:
Plan to Share IPD: No